CLINICAL TRIAL: NCT02705014
Title: Efficacy of Pulsatile GnRH Therapy on Male Patients With Pituitary Stalk Interruption Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, wuxueyan, professor,MD, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZS-997
Record Dates: First submitted 2016-02-22; First posted 2016-03-10 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Hypogonadotropic Hypogonadism
Keywords: pituitary stalk interruption syndrome; pulsatile GnRH therapy; hypogonadotropic hypogonadism; hypopituitarism
MeSH Terms: conditions — Hypogonadism; Hypopituitarism | interventions — Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment group (Experimental): patients were administered with pulsatile gonadotropin-releasing hormone (GnRH )therapy for 12 months at an interval of 90 minutes.The GnRH dosage was initially 10ug per pulse and was progressively adjusted to maintain serum testosterone levels at 6.94-17.35 nmol/L.
  Interventions: Drug: Gonadotropin-releasing Hormone

INTERVENTIONS:
Drug: Gonadotropin-releasing Hormone — A regimen of pulsatile GnRH (Fengyuan pharmaceutical company, Anhui province, China) administered subcutaneous via a portable infusion pump (Weichuang Medical Science Company, Shanghai city, China) at a 90-minute interval. The GnRH dosage was initially 10ug per pulse and was progressively adjusted to maintain serum testosterone levels at 6.94-17.35 nmol/L ( 200-500 ng/dL).
  Other Names: Gonadorelin

SUMMARY:
To investigate the hormone response of hypothalamic-pituitary-gonad axis and spermatogenesis in male pituitary stalk interruption syndrome patients by pulsatile GnRH therapy.

DETAILED DESCRIPTION:
To investigate the hormone response of hypothalamic-pituitary-gonad axis and spermatogenesis in male pituitary stalk interruption syndrome patients by pulsatile GnRH therapy. The hormonal response of the hypothalamic-pituitary-gonad axis was assessed after pulsatile GnRH replacement by measurement of serum T, LH and FSH. A standard seminal fluid analysis was performed in men who could produce an ejaculate.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or over male patients;
* Absent or incomplete puberty development;
* Serum testosterone values below 3.47 nmol/L by low or normal serum LH and FSH concentrations.
* at least two or more pituitary hormone deficiencies
* Brain MRI showed absent and thin pituitary stalk, or pituitary hypoplasia and/or ectopic posterior pituitary.

Exclusion Criteria:

* cryptorchidism history
* other causes of hypopituitarism or severe systemic disease

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Change of serum Luteinizing Hormone(LH) value | Baseline and at 1m,3m, 6m, 9m and 12m post treatment.
  Luteinizing hormone (LH) is measured using commercial kits by chemiluminescent method (ACS 180 Automatic Chemiluminescence System; Bayer). Reference range: 1.24-8.62 IU/L. Initial efficacy is evaluated based on the values of serum LH and serum total testosterone. If a subject's serum LH value below 1.5 IU/L and serum total testosterone value below 100 ng/dL at 3m post treatment, it is defined as failure to pulsatile GnRH treatment and continuous treatment is stopped. Otherwise, pulsatile GnRH treatment is continued.
Change of serum Follicle-Stimulating Hormone (FSH) value | Baseline and at 1m,3m, 6m, 9m and 12m post treatment.
  Follicle-stimulating hormone (FSH) are measured using commercial kits by chemiluminescent method (ACS 180 Automatic Chemiluminescence System; Bayer). Reference range: 1.27-19.26 IU/L.
Change of serum total testosterone value | Baseline and at 1m,3m, 6m, 9m and 12m post treatment.
  Total testosterone levels are measured using commercial kits by chemiluminescent method (ACS 180 Automatic Chemiluminescence System; Bayer). Reference range: 175-781 ng/dL.Initial efficacy is evaluated based on the values of serum LH and serum totaltestosterone. If a subject's serum LH value below 1.5 IU/L and serum total testosterone value below 100 ng/dL at 3m post treatment, it is defined as failure to pulsatile GnRH treatment and continuous treatment is stopped. Otherwise, pulsatile GnRH treatment is continued.

SECONDARY OUTCOMES:
Change of testicular volume | Baseline and at 1m,3m, 6m, 9m and 12m post treatment
  Testicular volumes are measured using Prader orchidometer. Prader orchidometer is a standard method to measure testicular volume. The normal range of testicular volume of each side in normal adult men is 15-25ml.
Change of sperm counts by routine semen analysis | Baseline and at 3m, 6m, 9m and 12m post treatment
  if a subject can produce an ejaculate, semen samples are collected by masturbation and analyzed according to the standard World Health Organization method.
the rate of impregnating subject's wife | at 3m, 6m, 9m and 12m post treatment
  For subjects who have sex partners, pregnancies are documented according to subjects' reports after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Xue-yan Wu, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shao WM, Bai WJ, Chen YM, Liu L, Wang YJ. [Micropump infusion of gonadorelin in the treatment of hypogonadotropic hypogonadism in patients with pituitary stalk interruption syndrome: cases analysis and literature review]. Beijing Da Xue Xue Bao Yi Xue Ban. 2014 Aug 18;46(4):642-5. Chinese. PMID 25131486
- [Derived] Zheng J, Mao J, Xu H, Wang X, Huang B, Liu Z, Cui M, Xiong S, Ma W, Min L, Kaiser UB, Nie M, Wu X. Pulsatile GnRH Therapy May Restore Hypothalamus-Pituitary-Testis Axis Function in Patients With Congenital Combined Pituitary Hormone Deficiency: A Prospective, Self-Controlled Trial. J Clin Endocrinol Metab. 2017 Jul 1;102(7):2291-2300. doi: 10.1210/jc.2016-3990. PMID 28368486